Study Title: Immersive virtual reality exposure for reducing preoperative anxiety in children – a randomized controlled trial

Central IRB Ref. No: HKCH-REC-2021-026

**NCT No: NCT07018999** 

**Document Title: Informed Consent Form** 

Version: 2.0

Version date: 14 August 2025

**Approved by:** Hospital Authority Central Institutional Review Board

(Central IRB), Hong Kong

**Initial approval version:** 31 August 2021 **Latest amendment approval:** 9 Sept 2025

**Note:** Study title is amended from 'Immersive virtual reality exposure for reducing *perioperative* anxiety in children – a randomized controlled trial' to Immersive virtual reality exposure for reducing *preoperative* anxiety in children – a randomized controlled trial' in year 2025 upon final submission of project and approved by Hospital Authority Central Institutional Review Board (Central IRB), Hong Kong

## **Study Title:**

Immersive virtual reality exposure for reducing preoperative anxiety in children – a randomized controlled trial

## Informed Consent Form (For subject's parent / legal guardian)

| (Please put a $\checkmark$ inside the appropriate check boxes $\square$ below.) |
|---|
| I hereby consent my child and I to participate in the research study. |
| I have read and understand this document. The study has been explained to me. I understand all the benefits and risks related to this study. I have opportunities to raise questions to the investigators and they have answered my questions to my satisfaction. I have collected sufficient information regarding this study. |
| If I have/my child has any physical or emotional discomfort as a result of participating in this study, the study investigators will treat me/my child, or will refer me/my child to receive treatment. Signing this informed consent form does not imply that my/my child's legal rights would be waived. |
| I understand that I can freely withdraw my/my child's consent on the participation of this study and is would not affect my/my child's present and future medical care. |
| I understand my/my child's identity will be kept confidential. I also authorize the research ethics committee and the regulatory authority(ies) to access my/my child's data for verification of clinical trial procedures and/or data, without violating my/my child's confidentiality, to the extent permitted by the applicable laws and regulations. |
| Data sharing I □ agree / □ do not agree that the research team can provide research results to online publicly available national/international databases to help clinicians, scientists and researchers understand the application of virtual reality in medical field. The results contained in the database will be made anonymous and thus not traceable to my/my child's record. |
| Use of data in scientific publication I □ agree / □ do not agree that clinical information and research results can be used in scientific publications. All direct identifiers shall be removed. Before the research investigators publish the results, the research investigators shall obtain approval from relevant regulatory bodies. If deemed necessary, the research investigators shall inform me about details of the publication. |

| Name of Participant | | |
|-------------------------------------------|-----------|------|
| Name of Parent / Legal Guardian | Signature | Date |
| (Specify Relationship with Participant) | | |
| Name of Research Investigator | Signature | Date |
| - | - | |
| Name of person taking consent | Signature | Date |
| (if different from Research Investigator) | | |
| Name of Witness (if applicable) | Signature | Date |

By signing a written informed consent form, I will be given a signed and dated copy of the consent form and information sheet for storage.